CLINICAL TRIAL: NCT02126228
Title: A Randomized Controlled Trial on Antibiotics Application For Low Infection-risked Elective Cesarean
Brief Title: no Antibiotics for Elective Cesarean With Low Risk of Infection
Status: Completed | Type: Observational
Sponsor: Fanzhen Hong (Other)
Responsible Party: Sponsor-Investigator, Fanzhen Hong, Obstetrics of 2nd Hopital, Shandong University
Organization: Shandong University (Other)
Other Study IDs: 2ndhsdu-ob
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Antibiotics , Elective Cesarean, China
Keywords: antibiotics, cesarean

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to discuss whether the parturients who underwent elective cesarean of such kind do not need prophylactic use of antibiotics and evaluate the risks and economic benefits involved.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean
* With normal temperature;
* No signs of infection;
* Normal degree of cleanliness in vaginal; .Normal amniotic fluid.

Exclusion Criteria:

* Failure of vaginal delivery and emergency cesarean;
* Premature rupture of membranes;
* Antibiotics having been applied to 3 days before cesarean;
* Having inflammation before cesarean: such as vaginitis, pelvic inflammatory disease, chorioamnionitis;
* Having infections in respiratory or urinary system before cesarean;
* Placenta previa or placental abruption;
* With medical and surgical complications;
* BMI ≥ 30kg/m2;
* Total blood loss more than 1000ml within 2 hours after cesarean

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: antibiotics group:202 none antibiotics group:212
Sampling Method: Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Temperature | 3days

SECONDARY OUTCOMES:
Postpartum hemorrhage volume estimates and Routine blood test. | 3days

OTHER OUTCOMES:
Observation of puerperal infection | 30days
  Incision healing;Intrauterine infection;Pelvic and abdominal infection;Infection of urinary system

CONTACTS AND LOCATIONS:
Overall Officials: YONGPING XU, MD.PhD, Study Director — Obstetrics of 2nd Hospital of Shandong University
Locations (1):
- 2nd Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Committee opinion no. 465: antimicrobial prophylaxis for cesarean delivery: timing of administration. Obstet Gynecol. 2010 Sep;116(3):791-792. doi: 10.1097/AOG.0b013e3181f68086. PMID 20733474